CLINICAL TRIAL: NCT01287039
Title: A 12-Month, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Reslizumab (3.0 mg/kg) in the Reduction of Clinical Asthma Exacerbations in Patients (12-75 Years of Age) With Eosinophilic Asthma
Brief Title: A Study to Evaluate the Efficacy and Safety of Reslizumab (3.0 mg/kg) in the Reduction of Clinical Asthma Exacerbations in Patients (12-75 Years of Age) With Eosinophilic Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C38072/3082
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — reslizumab; Antibodies, Monoclonal, Humanized

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered intravenously once every 4 weeks ( +-7 days) for a total of 13 doses.
  Interventions: Drug: Placebo
- Reslizumab 3.0 mg/kg (Experimental): Reslizumab 3.0 mg/kg administered intravenously once every 4 weeks ( +-7 days) for a total of 13 doses.
  Interventions: Drug: Reslizumab

INTERVENTIONS:
Drug: Reslizumab — Patients were administered intravenously over 15 to 30 minutes reslizumab at a dosage of 3.0 mg/kg at baseline and once every 4 weeks relative to baseline over 48 weeks for a total of 13 doses.
  Other Names: Cinquil; humanized monoclonal antibody; CEP-38072
  Arms: Reslizumab 3.0 mg/kg
Drug: Placebo — Matching placebo (20 mM sodium acetate, 7% sucrose), administered intravenously (iv) once every 4 weeks over 52 weeks, for a total of 13 doses administered. Each patient received a specific volume of placebo to match the volume of reslizumab on the basis of the patient's body weight.
  Arms: Placebo

SUMMARY:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy, safety, and immunogenicity of treatment with reslizumab in patients with eosinophilic asthma.

DETAILED DESCRIPTION:
Demonstrate the efficacy of reslizumab, at a dose of 3 mg/kg administered iv every 4 weeks over 12 months, as assessed by the reduction in frequency of clinical asthma exacerbations (CAEs) during 12 months.

An exacerbation event will be considered a CAE if the patient meets either or both of the criteria listed below and this is corroborated with at least 1 other measurement to indicate the worsening of clinical signs and symptoms of asthma:

* use of systemic, or an increase in the use of inhaled, corticosteroid treatment for 3 or more days
* asthma-related emergency treatment The above criteria must be corroborated with at least 1 other measurement to indicate worsening in the clinical signs and symptoms of asthma.

ELIGIBILITY:
Inclusion Criteria:

* The patient is male or female, 12 through 75 years of age, with a previous diagnosis of asthma.
* The patient has had at least 1 asthma exacerbation requiring oral, intramuscular (im), or intravenous (iv) corticosteroid use for at least 3 days over the past 12 months before screening.
* The patient has a current blood eosinophil level of at least 400/μl.
* The patient has airway reversibility of at least 12% to beta-agonist administration.
* The patient has an ACQ score of at least 1.5 at the screening and baseline (before the 1st dose of study drug) visits.
* The patient is taking inhaled fluticasone at a dosage of at least 440 μg, or equivalent, daily. Chronic oral corticosteroid use (no more than 10 mg/day prednisone or equivalent) is allowed. If a patient is on a stable dose, eg, 2 weeks or more of oral corticosteroid treatment at the time of study enrollment, the patient must remain on this dose throughout the study. The patient's baseline asthma therapy regimen (including but not limited to inhaled corticosteroids, oral corticosteroids up to a maximum of 10 mg of prednisone daily or equivalent, leukotriene antagonists, 5-lipooxygenase inhibitors, or cromolyn) must be stable for 30 days prior to screening and baseline, and must continue without dosage changes throughout study.
* All female patients must be surgically sterile, 2 years postmenopausal, or must have a negative pregnancy test ß-human chorionic gonadotropin [ß-HCG]) at screening (serum) and baseline (urine).
* Female patients of childbearing potential (not surgically sterile or 2 years postmenopausal), must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study.
* Written informed consent is obtained. Patients 12 through 17 years old must provide assent.
* The patient is in reasonable health (except for diagnosis of asthma) as judged by the investigator, and as determined by a medical history, medical examination, ECG evaluation (at screening), serum chemistry, hematology, and urinalysis.

  * Other criteria apply; please contact the investigator for more information.

Exclusion Criteria:

* The patient has a clinically meaningful co-morbidity that would interfere with the study schedule or procedures, or compromise the patient's safety.
* The patient has known hypereosinophilic syndrome.
* The patient has another confounding underlying lung disorder (eg, chronic obstructive pulmonary disease, pulmonary fibrosis, or lung cancer). Patients with pulmonary conditions with symptoms of asthma and blood eosinophilia (eg, Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis) will also be excluded.
* The patient is a current smoker (ie, has smoked within the last 6 months prior to screening).
* The patient is using systemic immunosuppressive or immunomodulating or other biologic agents (including, but not limited to, anti-IgE mAb, methotrexate, cyclosporin, interferon-α, or anti-tumor necrosis factor [anti TNF] mAb) within 6 months prior to screening.
* The patient has previously received an anti-hIL-5 monoclonal antibody (eg, reslizumab, mepolizumab, or benralizumab).
* The patient has any aggravating medical factors that are inadequately controlled (eg, rhinitis, gastroesophageal reflux disease, and uncontrolled diabetes).
* The patient has participated in any investigative drug or device study within 30 days prior to screening.
* The patient has participated in any investigative biologics study within 6 months prior to screening.
* Female patients who are pregnant, nursing, or, if of childbearing potential, and not using a medically accepted, effective method of birth control (eg, barrier method with spermicide, abstinence, IUD, or steroidal contraceptive [oral, transdermal, implanted, and injected]) are excluded from this study. NOTE: Partner sterility alone is not considered an acceptable form of birth control.

  * Other criteria apply; please contact the investigator for more information.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (128):
- United States (26):
  - Teva Investigational Site 58, Scottsdale, Arizona
  - Teva Investigational Site 61, Los Angeles, California
  - Teva Investigational Site 37, Orange, California
  - Teva Investigational Site 56, San Diego, California
  - Teva Investigational Site 34, Colorado Springs, Colorado
  - Teva Investigational Site 52, DeBary, Florida
  - Teva Investigational Site 55, Miami, Florida
  - Teva Investigational Site 18, Valrico, Florida
  - Teva Investigational Site 49, Lexington, Kentucky
  - Teva Investigational Site 65, Louisville, Kentucky
  - Teva Investigational Site 51, Boston, Massachusetts
  - Teva Investigational Site 74, St Louis, Missouri
  - Teva Investigational Site 35, Missoula, Montana
  - Teva Investigational Site 64, Boys Town, Nebraska
  - Teva Investigational Site 68, Rochester, New York
  - Teva Investigational Site 60, The Bronx, New York
  - Teva Investigational Site 30, Winston-Salem, North Carolina
  - Teva Investigational Site 31, Cincinnati, Ohio
  - Teva Investigational Site 62, Columbus, Ohio
  - Teva Investigational Site 50, Oklahoma City, Oklahoma
  - Teva Investigational Site 66, Altoona, Pennsylvania
  - Teva Investigational Site 32, Nashville, Tennessee
  - Teva Investigational Site 63, Boerne, Texas
  - Teva Investigational Site 72, Houston, Texas
  - Teva Investigational Site 38, Richmond, Virginia
  - Teva Investigational Site 33, Madison, Wisconsin
- Australia (5):
  - Teva Investigational Site 643, Nedlands, Western Australia
  - Teva Investigational Site 641, Clayton
  - Teva Investigational Site 644, Daw Park
  - Teva Investigational Site 642, Frankston
  - Teva Investigational Site 645, Liverpool
- Belgium (5):
  - Teva Investigational Site 261, Brussels
  - Teva Investigational Site 264, Brussels
  - Teva Investigational Site 260, Ghent
  - Teva Investigational Site 262, Jambes
  - Teva Investigational Site 263, Liège
- Chile (7):
  - Teva Investigational Site 160, Rancagua
  - Teva Investigational Site 163, Santiago
  - Teva Investigational Site 164, Santiago
  - Teva Investigational Site 165, Santiago
  - Teva Investigational Site 161, Temuco
  - Teva Investigational Site 162, Valdivia
  - Teva Investigational Site 166, Valparaíso
- Colombia (4):
  - Teva Investigational Site 181, Bogotá
  - Teva Investigational Site 185, Bogotá
  - Teva Investigational Site 182, Cali
  - Teva Investigational Site 180, Floridablanca
- Czechia (7):
  - Teva Investigational Site 287, Brno
  - Teva Investigational Site 284, Břeclav
  - Teva Investigational Site 286, Liberec
  - Teva Investigational Site 280, Olomouc
  - Teva Investigational Site 281, Olomouc
  - Teva Investigational Site 285, Olomouc
  - Teva Investigational Site 283, Tábor
- Denmark (2):
  - Teva Investigational Site 301, Hvidovre
  - Teva Investigational Site 300, Odense
- Hungary (5):
  - Teva Investigational Site 401, Balassagyarmat
  - Teva Investigational Site 400, Miskolc
  - Teva Investigational Site 404, Mosonmagyaróvár
  - Teva Investigational Site 403, Sopron
  - Teva Investigational Site 405, Törökbálint
- Israel (13):
  - Teva Investigational Site 423, Ashkelon
  - Teva Investigational Site 430, Beersheba
  - Teva Investigational Site 431, Haifa
  - Teva Investigational Site 432, Haifa
  - Teva Investigational Site 425, Jerusalem
  - Teva Investigational Site 428, Jerusalem
  - Teva Investigational Site 429, Jerusalem
  - Teva Investigational Site 426, Kfar Saba
  - Teva Investigational Site 422, Petah Tikva
  - Teva Investigational Site 427, Ramat Gan
  - Teva Investigational Site 433, Ramat Gan
  - Teva Investigational Site 421, Rehovot
  - Teva Investigational Site 420, Tel Aviv
- Malaysia (6):
  - Teva Investigational Site 705, Batu Caves
  - Teva Investigational Site 701, George Town
  - Teva Investigational Site 700, Kuala Lumpur
  - Teva Investigational Site 702, Kuala Lumpur
  - Teva Investigational Site 703, Kuantan
  - Teva Investigational Site 704, Taiping
- New Zealand (7):
  - Teva Investigational Site 723, Auckland
  - Teva Investigational Site 722, Christchurch
  - Teva Investigational Site 726, Christchurch
  - Teva Investigational Site 724, Dunedin
  - Teva Investigational Site 727, Hamilton
  - Teva Investigational Site 720, Tauranga
  - Teva Investigational Site 721, Wellington
- Philippines (6):
  - Teva Investigational Site 744, Governor Mangubat Drive, Dasma
  - Teva Investigational Site 742, Manila
  - Teva Investigational Site 740, Quezon City
  - Teva Investigational Site 741, Quezon City
  - Teva Investigational Site 743, Quezon City
  - Teva Investigational Site 745, Quezon City
- Poland (7):
  - Teva Investigational Site 507, Bialystok
  - Teva Investigational Site 509, Bydgoszcz
  - Teva Investigational Site 501, Bystra
  - Teva Investigational Site 500, Ostrów Wielkopolski
  - Teva Investigational Site 511, Poznan
  - Teva Investigational Site 502, Sopot
  - Teva Investigational Site 504, Tarnów
- Russia (9):
  - Teva Investigational Site 545, Barnaul
  - Teva Investigational Site 551, Kazan'
  - Teva Investigational Site 549, Kemerovo
  - Teva Investigational Site 550, Nizhny Novgorod
  - Teva Investigational Site 553, Novosibirsk
  - Teva Investigational Site 555, Novosibirsk
  - Teva Investigational Site 542, Saint Petersburg
  - Teva Investigational Site 552, Tomsk
  - Teva Investigational Site 546, Yaroslavl
- South Africa (10):
  - Teva Investigational Site 581, Cape Town
  - Teva Investigational Site 584, Cape Town
  - Teva Investigational Site 586, Cape Town
  - Teva Investigational Site 587, Centurion
  - Teva Investigational Site 582, Durban
  - Teva Investigational Site 585, Durban
  - Teva Investigational Site 580, Johannesburg
  - Teva Investigational Site 589, Johannesburg
  - Teva Investigational Site 583, Pretoria
  - Teva Investigational Site 588, Pretoria
- Sweden (4):
  - Teva Investigational Site 602, Gothenburg
  - Teva Investigational Site 604, Gothenburg
  - Teva Investigational Site 603, Linköping
  - Teva Investigational Site 601, Malmo
- Thailand (5):
  - Teva Investigational Site 780, Bangkok
  - Teva Investigational Site 782, Bangkok
  - Teva Investigational Site 783, Bangkok
  - Teva Investigational Site 781, Muang
  - Teva Investigational Site 784, Nakhon Ratchasima

REFERENCES:
- [Derived] Nair P, Bardin P, Humbert M, Murphy KR, Hickey L, Garin M, Vanlandingham R, Chanez P. Efficacy of Intravenous Reslizumab in Oral Corticosteroid-Dependent Asthma. J Allergy Clin Immunol Pract. 2020 Feb;8(2):555-564. doi: 10.1016/j.jaip.2019.09.036. Epub 2019 Oct 15. PMID 31626990
- [Derived] Carr WW, McDonald M, Meizlik P. Effect of intravenously administered reslizumab on spirometric lung age in patients with moderate-to-severe eosinophilic asthma. Allergy Asthma Proc. 2019 Jul 1;40(4):240-249. doi: 10.2500/aap.2019.40.4225. PMID 31262379
- [Derived] Han S, Kim S, Kim H, Suh HS. Cost-utility analysis of reslizumab for patients with severe eosinophilic asthma inadequately controlled with high-dose inhaled corticosteroids and long-acting beta2-agonists in South Korea. Curr Med Res Opin. 2019 Sep;35(9):1597-1605. doi: 10.1080/03007995.2019.1605159. Epub 2019 May 16. PMID 30964365
- [Derived] Bateman ED, Djukanovic R, Castro M, Canvin J, Germinaro M, Noble R, Garin M, Buhl R. Predicting Responders to Reslizumab after 16 Weeks of Treatment Using an Algorithm Derived from Clinical Studies of Patients with Severe Eosinophilic Asthma. Am J Respir Crit Care Med. 2019 Feb 15;199(4):489-495. doi: 10.1164/rccm.201708-1668OC. PMID 30346831
- [Derived] Weinstein SF, Katial RK, Bardin P, Korn S, McDonald M, Garin M, Bateman ED, Hoyte FCL, Germinaro M. Effects of Reslizumab on Asthma Outcomes in a Subgroup of Eosinophilic Asthma Patients with Self-Reported Chronic Rhinosinusitis with Nasal Polyps. J Allergy Clin Immunol Pract. 2019 Feb;7(2):589-596.e3. doi: 10.1016/j.jaip.2018.08.021. Epub 2018 Sep 5. PMID 30193936
- [Derived] Brusselle G, Germinaro M, Weiss S, Zangrilli J. Reslizumab in patients with inadequately controlled late-onset asthma and elevated blood eosinophils. Pulm Pharmacol Ther. 2017 Apr;43:39-45. doi: 10.1016/j.pupt.2017.01.011. Epub 2017 Jan 31. PMID 28159511
- [Derived] Castro M, Zangrilli J, Wechsler ME, Bateman ED, Brusselle GG, Bardin P, Murphy K, Maspero JF, O'Brien C, Korn S. Reslizumab for inadequately controlled asthma with elevated blood eosinophil counts: results from two multicentre, parallel, double-blind, randomised, placebo-controlled, phase 3 trials. Lancet Respir Med. 2015 May;3(5):355-66. doi: 10.1016/S2213-2600(15)00042-9. Epub 2015 Feb 23. PMID 25736990

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1486 patients were screened at 121 centers. Of the 1486 patients screened, 489 patients with asthma and blood eosinophils ≥400/ μL at 102 centers in 17 countries were randomly assigned to double-blind treatment.
Pre-assignment Details: 997 of 1486 screened patients were not randomized: 888 were excluded on the basis of not meeting inclusion criteria, 23 withdrew consent, 17 had an adverse event during the screening period, 12 met an exclusion criterion, 7 were lost to follow-up and 50 were excluded for other reasons. One placebo patient was randomized but not treated.
Period: Overall Study
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Started | 244 | 245
Completed | 215 | 218
Not Completed | 29 | 27
Not completed — Noncompliance with study procedures | 0 | 1
Not completed — Change of location/residence | 0 | 3
Not completed — Elective surgery | 0 | 1
Not completed — Protocol Violation | 2 | 3
Not completed — Excluded medication taken | 1 | 0
Not completed — Noncompliance with study medication | 0 | 1
Not completed — Problem with travel | 0 | 1
Not completed — Death | 1 | 0
Not completed — Change of residence | 1 | 0
Not completed — Adverse Event | 7 | 4
Not completed — Withdrawal by Subject | 14 | 11
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Population: Randomized set
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Reslizumab 3.0 mg/kg | Total
Number analyzed (Participants) | 244 | 245 | 489
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (14.83) | 46.6 (13.82) | 46.6 (14.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 142 | 303
  Male | 83 | 103 | 186
Race/Ethnicity, Customized [Number; unit: participants]
  White | 182 | 173 | 355
  Black | 20 | 14 | 34
  Asian | 33 | 50 | 83
  American Indian or Alaskan Native | 0 | 0 | 0
  Pacific Islander | 0 | 1 | 1
  Other | 9 | 7 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic and non-Latino | 223 | 216 | 439
  Hispanic or Latino | 21 | 28 | 49
  Unknown | 0 | 1 | 1
Weight [Mean (Standard Deviation); unit: kg] | 76.5 (18.71) | 75.6 (19.05) | 76.0 (18.87)
Height [Mean (Standard Deviation); unit: cm] | 165.0 (9.74) | 164.9 (10.42) | 164.9 (10.07)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (6.16) | 27.7 (6.26) | 27.9 (6.20)
Oral Glucocorticosteroid (OCS) Use at Baseline [Number; unit: participants] — Oral glucocorticosteroid (OCS) use at baseline was a stratification factor. Values input by the investigator into the interactive response technology (IRT) were used during randomization. However, 6 patients in the placebo group and 22 patients in the reslizumab group were misclassified in IRT as having used oral glucocorticosteroids at baseline according to the case report form.
  participants
    OCS - Yes | 46 | 46 | 92
    OCS - No | 198 | 199 | 397
Asthma Exacerbations In Previous 12 Months [Mean (Standard Deviation); unit: exacerbations] | 2.1 (2.31) | 1.9 (1.63) | 2.0 (2.00)
Forced Expiratory Volume in 1 Second [Mean (Standard Deviation); unit: liters] | 1.928 (0.7908) | 1.894 (0.7258) | 1.911 (0.7583)
Asthma Control Questionnaire (ACQ) Overall Score [Mean (Standard Deviation); unit: units on a scale] — The ACQ is a 7-item instrument that measures asthma control (Juniper et al 1999). Six questions are self-assessments; the seventh item, completed by a member of the study staff, is the result of the patient's FEV1 measurement. Each item has 7 possible answers on a scale of 0 to 6, and the overall score is the mean of all responses. A higher score is an indication of poorer asthma control.
  units on a scale | 2.763 (0.8782) | 2.657 (0.8541) | 2.710 (0.867)
Asthma Quality of Life Questionnaire (AQLQ) [Mean (Standard Deviation); unit: units on a scale] — The AQLQ is a 32-item instrument administered as a self-assessment (Juniper et al 1992). The questionnaire is divided into 4 domains: activity limitation, symptoms, emotional function, and environmental stimuli. Patients were asked to recall their experiences during the last 2 weeks and to respond to each question on a 7-point scale (1=severe impairment, 7=no impairment). The overall AQLQ score is the mean of all 32 responses.
  units on a scale | 4.159 (1.0883) | 4.303 (1.1208) | 4.231 (1.1059)
Asthma Symptom Utility Index (ASUI) [Mean (Standard Deviation); unit: units on a scale] — The ASUI is an 11-item instrument designed to assess the frequency and severity of asthma symptoms and side effects, weighted by patient preferences (Revicki et al 1998). ASUI is a utility score that ranges from 0 to 1, with higher values indicating better asthma control.
  units on a scale | 0.613 (0.2029) | 0.633 (0.1938) | 0.623 (0.1984)
Number of Short-Acting Beta-Agonist Puffs (SABA) Daily [Mean (Standard Deviation); unit: puffs/day] — Based on patient-reported total number of SABA puffs over the past 3 days.
  puffs/day | 2.7 (3.18) | 2.4 (2.82) | 2.6 (3.01)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Clinical Asthma Exacerbations (CAEs) During 12 Months of Treatment
Description: An exacerbation event was considered a CAE if the patient met either or both of the criteria listed below and this was corroborated with at least 1 other measurement to indicate the worsening of clinical signs and symptoms of asthma:
  * use of systemic, or an increase in the use of inhaled, corticosteroid treatment for 3 or more days; or an increased 2 or more fold for at least 3 or more days for patient's already on corticosteroids.
  * asthma-related emergency treatment, such as an unscheduled visit to the physician's office or emergency room for nebulizer treatment or other urgent treatment to prevent worsening of asthma symptoms, or an asthma-related hospitalization CAEs were adjudicated by committee to assure consistency.
  Adjusted CAE rate and confidence intervals were based on Negative Binomial regression model adjusted for stratification factors.
  Results are offered as adjusted means.
Time Frame: Day 1 to Week 52
Population: Randomized set
Measure: Mean (95% Confidence Interval); unit: CAEs in 52 weeks
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 244 | 245
CAEs in 52 weeks | 1.804 [1.372 to 2.372] | 0.904 [0.678 to 1.205]
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; The frequency of CAEs was analyzed using the generalized linear model (GLM) for data from the negative binomial distributions that is commonly referred to as the negative binomial (NB) regression model. The primary NB model included the treatment group and randomization stratification factors as model factors and the logarithm of follow up time excluding the summed duration of exacerbations in the treatment period as an offset variable; Test type: Superiority or Other; p < 0.0001, Chi-squared — The treatment effect was tested using the likelihood based Chi-square test at the 0.05 significance level; CAE rate ratio (reslizumab vs placebo) = 0.5010, 95% CI 2-sided [0.3726 to 0.6737]

2. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Over 16 Weeks Using Mixed Model for Repeated Measures
Description: FEV1 is a standard measurement of air movement in the lungs of patients with asthma obtained from pulmonary function tests. It is the volume of air expired in the first second of a forced expiration using a spirometer. Positive change from baseline scores indicate improvement in asthma control.
  The during treatment (Weeks 4, 8, 12 and 16) average FEV1 was estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12 and 16
Population: Randomized set, including participants who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 241 | 243
liters | 0.110 (0.031) | 0.248 (0.030)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; For each week and overall change, inferential statistics were from mixed model repeated measures (MMRM) with treatment, visit, treatment by visit interaction, region, oral glucocorticosteroids use at enrollment and sex as fixed factors, and covariates for height and baseline value and patient as a random effect. Unstructured covariance structure was assumed for the repeated measures; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures; Mean Difference (Net) = 0.137, 95% CI 2-sided [0.076 to 0.198], Standard Error of Mean 0.0311

3. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (AQLQ) to Week 16
Description: The AQLQ is a 32-item instrument administered as a self-assessment (Juniper et al 1992). The questionnaire is divided into 4 domains: activity limitation, symptoms, emotional function, and environmental stimuli. Patients were asked to recall their experiences during the last 2 weeks and to respond to each question on a 7-point scale (1=severe impairment, 7=no impairment). The overall AQLQ score is the mean of all 32 responses. Five of the activity questions were "patient-specific," which means that each patient identified and scored 5 activities in which the patient was limited by asthma; these 5 activities were identified at the first visit and retained for all subsequent follow-up visits.
  Positive change from baseline scores indicate improvement in quality of life.
Time Frame: Day 1 (baseline, pre-dose), Week 16
Population: Randomized set of patients with assessments at both timepoints
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 229 | 228
units on a scale | 0.695 (0.088) | 0.933 (0.088)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0143, Mixed model repeated measures; Mean Difference (Final Values) = 0.238, 95% CI 2-sided [0.048 to 0.428], Standard Error of Mean 0.0967

4. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) Over 16 Weeks Using Mixed Model for Repeated Measures
Description: The ACQ is a 7-item instrument that measures asthma control (Juniper et al 1999). Six questions are self-assessments; the seventh item, completed by a member of the study staff, is the result of the patient's FEV1 measurement. Each item has 7 possible answers on a scale of 0 to 6, and the total score is the mean of all responses (the total scale is therefore 0-6). A higher score is an indication of poorer asthma control. The during treatment (Weeks 4, 8, 12 and 16) average ACQ was estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
  Negative change from baseline scores indicate improvement in asthma control.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16
Population: Randomized set, including participants who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 241 | 242
units on a scale | -0.676 (0.066) | -0.941 (0.065)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0001, Mixed model repeated measures; Mean Difference (Final Values) = -0.266, 95% CI 2-sided [-0.399 to -0.132], Standard Error of Mean 0.0681

5. Secondary Outcome: Kaplan-Meier Estimates for Time to First Clinical Asthma Exacerbation (CAE)
Description: An exacerbation event was considered a CAE if the patient met either or both of the criteria listed below and this was corroborated with at least 1 other measurement to indicate the worsening of clinical signs and symptoms of asthma:
  * use of systemic, or an increase in the use of inhaled, corticosteroid treatment for 3 or more days; or an increased 2 or more fold for at least 3 or more days for patient's already on corticosteroids.
  * asthma-related emergency treatment, such as an unscheduled visit to the physician's office or emergency room for nebulizer treatment or other urgent treatment to prevent worsening of asthma symptoms, or an asthma-related hospitalization.
  CAEs were adjudicated by committee to assure consistency. The distributions were compared by a log rank test stratified by baseline usage of oral corticosteroid (yes or no) and geographical region (US or other).
Time Frame: Day 1 to Day 478 (longest treatment time plus 2 weeks)
Population: Randomized set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 244 | 245
weeks | 34.9 [23.3 to NA] — Insufficient data to estimate time | NA [NA to NA] — Insufficient data to estimate time
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; Kaplan-Meier estimate of probability (5) of not experiencing a CAE by week 52. The first CAEs for each patient occurring after randomization and up to 2 weeks after the end of treatment period were analyzed. Patients without a CAE within this time frame were censored at two weeks after the treatment completion date or study discontinuation, whichever came first; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Stratified by baseline usage of oral corticosteroid (yes or no) and geographical region (US or other); Cox Proportional Hazard = 0.575, 95% CI 2-sided [0.440 to 0.750] — Reslizumab vs placebo

6. Secondary Outcome: Change From Baseline in Asthma Symptom Utility Index (ASUI) Over 16 Weeks Using Mixed Model for Repeated Measures
Description: The ASUI is an 11-item instrument designed to assess the frequency and severity of asthma symptoms and side effects, weighted by patient preferences (Revicki et al 1998). ASUI is a utility score that ranges from 0 to 1, with higher values indicating better asthma control; info obtained from questionnaire about asthma symptoms.
  The during treatment (Weeks 4, 8, 12 and 16) average ASUI was estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
  Positive change from baseline values indicate improvement in asthma symptoms. Information was obtained from questionnaire about asthma symptoms.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16
Population: Randomized set, including participants who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 238 | 238
units on a scale | 0.109 (0.012) | 0.167 (0.188)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; For each week, inferential statistics were from mixed model repeated measures (MMRM) with treatment, visit, treatment by visit interaction, region, oral glucocorticosteroids use at enrollment as fixed factor, and covariate baseline value and patient as a random effect. Unstructured covariance structure was assumed for the repeated measures; Test type: Superiority or Other; p < 0.0001, Mixed model repeated measures; Median Difference (Final Values) = 0.058, 95% CI 2-sided [0.034 to 0.083], Standard Error of Mean 0.0125

7. Secondary Outcome: Change From Baseline in Short-Acting Beta-Agonist (SABA) Use Over 16 Weeks Using Mixed Model for Repeated Measures
Description: SABA are used for quick relief of asthma symptoms. To measure SABA use, at each clinical visit patients were asked to recall their usage of SABA therapy within the last 3 days of the scheduled visit. If usage was confirmed, the number of puffs used was recorded. For the purpose of summaries, an average daily usage was evaluated by dividing the total number of puffs recorded over 3 days by 3.
  The during treatment (Weeks 4, 8, 12 and 16) SABA use was estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
  Negative change from baseline scores indicate improvement in asthma control.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16
Population: Randomized set of participants with assessments within the timeframe
Measure: Least Squares Mean (Standard Error); unit: puffs/day
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 238 | 240
puffs/day | -0.36 (0.158) | -0.64 (0.156)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; Inferential statistics were from mixed model repeated measures (MMRM) with treatment, visit, treatment by visit interaction, region, OCS use at enrollment as fixed factors, and covariate for baseline value and patient as a random effect. Unstructured covariance structure was assumed for the repeated measures; Test type: Superiority or Other; p = 0.0919, Mixed model repeated measures; Mean Difference (Final Values) = -0.276, 95% CI 2-sided [-0.597 to 0.045], Standard Error of Mean 0.1632

8. Secondary Outcome: Change From Baseline in Blood Eosinophil Count Over 16 Weeks and 52 Weeks Using Mixed Model for Repeated Measures
Description: Blood eosinophil counts were measured using a standard complete blood count (CBC) with differential blood test at each scheduled visit, and from all patients experiencing a serious adverse event, an adverse event leading to withdrawal, or an exacerbation of asthma symptoms.
  The during treatment average eosinophil counts were estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
  Negative change from baseline values correlate to reduced asthma severity.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 or early withdrawal
Population: Randomized set of participants with assessments within timeframe
Measure: Least Squares Mean (Standard Error); unit: 10^9 blood eosinophil/L
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 241 | 243
10^9 blood eosinophil/L
  Over first 16 weeks | -0.118 (0.0232) | -0.584 (0.0230)
  Over 52 weeks | -0.127 (0.0168) | -0.582 (0.0167)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; Eosinophil Count Over 16 Weeks Inferential statistics were from mixed model repeated measures (MMRM) with treatment, visit, treatment by visit interaction, region, oral glucocorticosteroids use at enrollment as fixed factor, and covariate baseline value and patient as a random effect. Unstructured covariance structure was assumed for the repeated measures; Test type: Superiority or Other; p < 0.0001, Mixed model repeated measures; Mean Difference (Final Values) = -0.466, 95% CI 2-sided [-0.514 to -0.418], Standard Error of Mean 0.0244
Statistical Analysis 2: Comparison: Placebo vs Reslizumab 3.0 mg/kg; Eosinophil Count Over 52 Weeks Inferential statistics were from mixed model repeated measures (MMRM) with treatment, visit, treatment by visit interaction, region, oral glucocorticosteroids use at enrollment as fixed factor, and covariate baseline value and patient as a random effect. Unstructured covariance structure was assumed for the repeated measures; Test type: Superiority or Other; p < 0.0001, Mixed model repeated measures; Mean Difference (Final Values) = -0.455, 95% CI 2-sided [-0.491 to -0.419], Standard Error of Mean 0.0182

9. Secondary Outcome: Participants With Treatment-Emergent Adverse Events
Description: An adverse event was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an inability to carry out usual activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 (post-dose) to Week 65. The last postbaseline value for approximately 20 patients in each
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 243 | 245
participants
  At least 1 AE | 206 | 197
  Mild severity AE | 41 | 68
  Moderate severity AE | 133 | 107
  Severe AE | 32 | 22
  Treatment-related AE | 36 | 36
  Treatment-related mild AE | 23 | 24
  Treatment-related moderate AE | 13 | 9
  Treatment-related severe AE | 0 | 3
  AE causing patient discontinuation | 8 | 4
  Serious AE | 34 | 24
  Deaths | 1 | 0

10. Primary Outcome: Frequency of Each of the Two Criteria for Clinical Asthma Exacerbations (CAEs)
Description: An exacerbation event was considered a CAE if the patient met either or both of the criteria listed below and this was corroborated with at least 1 other measurement to indicate the worsening of clinical signs and symptoms of asthma:
  * use of systemic, or an increase in the use of inhaled, corticosteroid treatment for 3 or more days; or an increased 2 or more fold for at least 3 or more days for patient's already on corticosteroids.
  * asthma-related emergency treatment, such as an unscheduled visit to the physician's office or emergency room for nebulizer treatment or other urgent treatment to prevent worsening of asthma symptoms, or an asthma-related hospitalization.
  CAEs were adjudicated by committee to assure consistency. Adjusted CAE rate and confidence intervals for the two criteria were based on Negative Binomial regression model adjusted for stratification factors.
  Results are offered as adjusted means.
Time Frame: Day 1 to Week 52
Population: Randomized set
Measure: Mean (95% Confidence Interval); unit: CAEs in 52 weeks
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 244 | 245
CAEs in 52 weeks
  Requiring systemic corticosterioids >3 days | 1.604 [1.195 to 2.152] | 0.722 [0.528 to 0.986]
  Requiring hospitalization or ER visit | 0.207 [0.107 to 0.400] | 0.137 [0.068 to 0.274]
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; CAE Due to Requiring Systemic Corticosteroids The frequency of CAEs was analyzed using the generalized linear model (GLM) for data from the negative binomial distributions that is commonly referred to as the negative binomial (NB) regression model. The primary NB model included the treatment group and randomization stratification factors as model factors and the logarithm of follow up time excluding the summed duration of exacerbations in the treatment period as an offset variable; Test type: Superiority or Other; p < 0.0001, Chi-squared — The treatment effect was tested using the likelihood based Chi-square test at the 0.05 significance level; CAE rate ratio (reslizumab vs placebo) = 0.4499, 95% CI 2-sided [0.3255 to 0.6220]
Statistical Analysis 2: Comparison: Placebo vs Reslizumab 3.0 mg/kg; CAE Due to Hospitalization or ER visit The frequency of CAEs was analyzed using the generalized linear model (GLM) for data from the negative binomial distributions that is commonly referred to as the negative binomial (NB) regression model. The primary NB model included the treatment group and randomization stratification factors as model factors and the logarithm of follow up time excluding the summed duration of exacerbations in the treatment period as an offset variable; Test type: Superiority or Other; p = 0.2572, Chi-squared — The treatment effect was tested using the likelihood based Chi-square test at the 0.05 significance level; CAE rate ratio (reslizumab vs placebo) = 0.6595, 95% CI 2-sided [0.3210 to 1.3550]

11. Secondary Outcome: Participants With Treatment-Emergent Potentially Clinically Significant (PCS) Abnormal Lab Values
Description: Data represents participants with potentially clinically significant (PCS) abnormal serum chemistry, hematology, and urinalysis values.
  Significance criteria:
  * Blood urea nitrogen: >=10.71 mmol/L
  * Uric acid: M>=625, F>=506 μmol/L
  * Aspartate aminotransferase: >=3*upper limit of normal (ULN). Normal range is 10-43 U/L
  * Alanine aminotransferase: >=3*ULN. Normal range is 10-40 U/L
  * GGT = gamma-glutamyl transpeptidase: >= 3*ULN. Normal range is 5-49 U/L.
  * Bilirubin: >=34.2 μmol/L
  * White blood cells: <=3.0 or >20 10^9/L
  * Hemoglobin: M<=115, F<=95 g/dL
  * Hematocrit: M<0.37, F<0.32 L/L
  * Neutrophils: <=1.0 10^9/L
  * Eosinophils: >10.0 %
  * Platelets: <75 or >=700 10^9/L
  * Urinalysis: blood, glucose, ketones and total protein: >=2 unit increase from baseline
Time Frame: Week 4 to Week 65. The last postbaseline value for approximately 20 patients in each
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 243 | 245
participants
  Blood urea nitrogen | 9 | 8
  Uric acid | 9 | 6
  Aspartate aminotransferase | 1 | 1
  Alanine aminotransferase | 3 | 5
  Gamma-glutamyl transpeptidase | 12 | 12
  Bilirubin | 2 | 1
  White blood cells - low | 6 | 6
  White blood cells - high | 5 | 3
  Hemoglobin | 7 | 4
  Hematocrit | 9 | 6
  Neutrophils | 8 | 6
  Eosinophils | 135 | 3
  Platelets - low | 1 | 2
  Platelets - high | 2 | 0
  Urinalysis - Blood (hemoglobin) | 32 | 21
  Urinalysis - Ketones | 4 | 5
  Urinalysis - Glucose | 11 | 14
  Urinalysis - Protein | 32 | 34

12. Secondary Outcome: Participants With Treatment-Emergent Potentially Clinically Significant (PCS) Vital Signs Values
Description: Data represents participants with potentially clinically significant (PCS) vital sign values.
  Significance criteria
  * Sitting pulse - high 12-17 yr: >100 and increase of >= 30 beats/minute (bpm)
  * Sitting pulse - low >=18 yr: <50 and decrease of >=30 bpm
  * Sitting pulse - high >=18 yr: >100 and increase of >=30 bpm
  * Sitting systolic blood pressure - low >=18 yr: <90 and decrease of >=30 mmHg
  * Sitting systolic blood pressure - high >=18 yr: >160 and increase of >=30 mmHg
  * Sitting diastolic blood pressure - low 12-17 yr: <55 and decrease of >=12 mmHg
  * Sitting diastolic blood pressure - low >=18 yr: <50 and decrease of >=12 mmHg
  * Sitting diastolic blood pressure - high >=18 yr: >100 and increase of >=12 mmHg
  * Respiratory rate >=18 yr: >24 and increase of >=10 breaths/minute
  * Body temperature - low 12-17 yr: <96.5° Fahrenheit or <35.8° Celsius
  * Body temp - low >=18 yr: <96.5° F or <35.8° C
  * Body temp - high >=18 yr: >100.5° Fahrenheit
Time Frame: Week 4 to Week 65. The last postbaseline value for approximately 20 patients in each
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 243 | 245
participants
  Sitting pulse - high 12-17 yr | 1 | 1
  Sitting pulse - low >=18 yr | 1 | 0
  Sitting pulse - high >=18 yr | 5 | 7
  Sitting systolic blood pressure - low >=18 yr | 2 | 5
  Sitting systolic blood pressure - high >=18 yr | 7 | 7
  Sitting diastolic blood pressure - low 12-17 yr | 1 | 0
  Sitting diastolic blood pressure - low >=18 yr | 0 | 1
  Sitting diastolic blood pressure - high >=18 yr | 10 | 5
  Respiratory rate >=18 yr | 3 | 2
  Body temperature - low 12-17 yr | 1 | 1
  Body temperature - low >=18 yr | 54 | 49
  Body temperature - high >=18 yr | 0 | 1

13. Secondary Outcome: Participants With a Positive Anti-Reslizumab Antibody Status During Study
Description: The immunogenicity of reslizumab was assessed by measuring for the presence of anti-reslizumab antibodies at baseline, weeks 16, 32, 48, and 52 or early withdrawal. Blood samples for anti-reslizumab antibodies assessment were also obtained from all patients (inside or outside of the US) experiencing a serious adverse event, an adverse event leading to withdrawal, or an exacerbation of asthma symptoms.
Time Frame: Weeks 16, 32, 48 and 52
Population: Safety analysis set. Immunogenicity for anti-reslizumab antibodies not reported for the placebo treatment arm.
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 0 | 245
participants |  | 8

ADVERSE EVENTS:
Time Frame: Day 1 to Day 464
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 34/243 | 24/245
Other Adverse Events (participants affected / at risk) | 184/243 | 165/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=243) | Reslizumab 3.0 mg/kg (N=245)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 2 (3) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningism (Nervous system disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0)
Status migrainosus (Nervous system disorders) | 1 (2) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 13 (28) | 11 (12)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=243) | Reslizumab 3.0 mg/kg (N=245)
Bronchitis (Infections and infestations) | 22 (31) | 13 (14)
Influenza (Infections and infestations) | 23 (32) | 17 (25)
Nasopharyngitis (Infections and infestations) | 33 (44) | 28 (45)
Pharyngitis (Infections and infestations) | 13 (13) | 10 (11)
Sinusitis (Infections and infestations) | 28 (48) | 21 (31)
Upper respiratory tract infection (Infections and infestations) | 32 (49) | 39 (50)
Urinary tract infection (Infections and infestations) | 10 (13) | 13 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 13 (15)
Dizziness (Nervous system disorders) | 13 (13) | 5 (7)
Headache (Nervous system disorders) | 30 (50) | 19 (31)
Asthma (Respiratory, thoracic and mediastinal disorders) | 123 (364) | 92 (192)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 11 (13)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 13 (17)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 13 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.